CLINICAL TRIAL: NCT03329157
Title: Rebuilding Bridges for Homeless Veterans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was planned but never formally commenced and PI moved institutions.
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 102317
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Housing Problems

STUDY DESIGN:
Intervention Model Description: Single group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rebuilding Bridges (Other): This is a one-group study and the group will receive the Rebuilding Bridges intervention
  Interventions: Other: Rebuilding Bridges

INTERVENTIONS:
Other: Rebuilding Bridges — Psychosocial intervention to help veterans re-engage with family members called Rebuilding Bridges, developed for this project.

SUMMARY:
Pilot study on an intervention called Rebuilding Bridges to help veterans re-engaged with loved ones.

DETAILED DESCRIPTION:
The objective of the proposed project is to examine the feasibility and acceptability of the Rebuilding Bridges intervention, which was designed to help homeless Veterans plan and implement steps to engage friends, family and other loved ones in their lives. The PI and his team will enroll approximately 25-30 Veterans. Veterans will be recruited via provider referral and via advertisements that will be placed in general clinical areas and desks at the Errera Center. The PI will work with the Veterans to create a detailed genogram of family, friends and other supporters in the Veteran's life. This will be followed by a meeting with each Veteran over the course of three 30-minute weekly sessions to help the Veteran identify and engage people listed in their genogram which the Veteran might want to form stronger relationships with. Veterans will also be asked to complete several measures and questionnaires such as housing information, employment, mental health and quality of life.

ELIGIBILITY:
Inclusion Criteria

1. Over 18 years old
2. Currently in a VA homeless program
3. Able to provide valid consent

Exclusion Criteria

1. Acute psychiatric decompensation requiring inpatient admission or emergency department services within the last month (suicidality, homicidally, mania, psychotic decompensation)
2. Has a conservator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Social Support | 2 years
  2-Way Social Support scale and the Multidimensional Scale of Perceived Social Support, which generates a total score from 1 to 7 with higher scores indicating greater social support

SECONDARY OUTCOMES:
Housing status | 2 years
  Nights stayed in own place and nights homeless in the past 60 days, which should total 60 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Tsai, PhD, Principal Investigator — VA Connecticut
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No